CLINICAL TRIAL: NCT02664038
Title: Cognitive Training in the Treatment of Alcohol Use Disorders in Older Veterans
Brief Title: Cognitive Training in the Treatment of AUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2017-R
Record Dates: First submitted 2016-01-14; First posted 2016-01-26 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder Cognitive Decline
Keywords: AUD; Neuropsychology; Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRT+IDC (Experimental): Cognitive Remediation Therapy for 13 weeks plus Individual Drug Counseling
  Interventions: Behavioral: Cognitive Remediation Training
- Computer Game Play+IDC (Active Comparator): Computer arcade games for 13 weeks plus Individual Drug Counseling
  Interventions: Behavioral: Cognitive Remediation Training

INTERVENTIONS:
Behavioral: Cognitive Remediation Training — Up to 65 hours of computer based cognitive training of attention, verbal and visual memory, verbal and visual working memory, and executive functions

SUMMARY:
Alcohol Use Disorders (AUDs) have a significant public health impact and are highly prevalent in Veterans. Alcohol related brain effects on neurocognition (attention, memory and executive function) reduce ability to benefit from current treatments. These cognitive impairments are especially common in the early phase of recovery, persist over years and get worse with age. Recent research suggests that cognitive remediation therapy (CRT) may improve attention, memory and executive function in other disorders, and the investigators just completed pilot study with AUD Veterans found significantly greater improvements for those receiving CRT. The proposed study examines AUD outcomes and neurocognitive improvements when CRT is combined with a standardized alcohol treatment. The investigators hypothesize that CRT will improve neurocognition and AUD outcomes more than standardized alcohol treatment alone. Findings will determine whether CRT augmentation can benefit Veterans with AUDs.

DETAILED DESCRIPTION:
This study aims to determine whether a combined intervention of cognitive remediation therapy (CRT) and Individual Drug Counseling (IDC) can benefit older Veterans in the initial phase of alcohol abuse treatment by improving abstinence outcomes and neurocognition. Substantial cognitive impairment is associated with alcohol use disorders (AUD), and becomes worse with years of use and the aging processes. In particular, Veterans entering treatment for AUD display cognitive deficits that may reduce their ability to benefit from treatment. While there is considerable variety in the severity and types of cognitive impairment found in newly recovering patients, problems with attention, learning and memory and executive function are common. Since treatment requires that the individual be able to sustain attention, remember what is learned, and apply it to recovery, impaired underlying cognitive processes make successful treatment less likely. Moreover, problems with executive functioning and other pre-frontal cognitive processes have been associated with decreased treatment retention and poorer AUD treatment outcomes. Although cognition can improve with sustained abstinence, it is during the early phase of recovery, when cognition is most impaired, that patients receive the most intensive treatment. AUD is a major cause of suffering and functional disability for older Veterans and a common co-morbidity with other physical and mental disorders. Finding more effective treatments of AUD remains a priority for VA healthcare.

The purpose of the proposed study is to learn whether CRT plus IDC, an evidence-based outpatient AUD treatment is more effective than a Game-Play Placebo plus IDC. Game-Play Placebo has been used to provide equipoise between conditions in other CRT studies and in a current CRT study with mTBI Veterans funded by DoD being conducted by the PI. The current study is a randomized controlled trial (RCT) with a target enrollment of 90 Veterans in the initial phase of AUD treatment. The study is sufficiently powered to allow us to fulfill the following aims and test their related hypotheses:

Specific Primary Aim # 1: To determine if CRT+IDC is more effective than Game-Play Placebo +IDC in decreasing alcohol use in older Veterans during the 3 month active intervention period.

Ho1: CRT+IDC will be more effective than Game-Play Placebo+IDC in reducing heavy drinking days and decreasing days of use as measured by Breathalyzer and Timeline Follow-back Method (TLFB) during the 90 days of active intervention.

Secondary Aim #1: To determine if CRT+IDC is more effective than Game-Play Placebo+ IDC in sustaining decreased alcohol use in older Veterans at the end of 6 months (3 months after the active intervention period).

Ho2: CRT+IDC will be more effective than Game-Play Placebo+IDC in reducing heavy drinking days and decreasing days of use as measured by Breathalyzer and Timeline Follow-back Method (TLFB) for the 30 days preceding 6 month follow-up.

Secondary Aim #2: To determine if the combination of CRT and IDC is more effective than game play placebo and IDC in improving neurocognitive functioning.

Ho3: Veterans receiving CRT+IDC will show greater improvement than Veterans receiving Game-Play Placebo+IDC at 3 month follow-up on a global index of neurocognitive function, and on an index of working memory and an index of executive function.

Ho4: Differential improvements in neurocognitive function will be sustained at 6 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled in VA AUD treatment as usual and Non-Veteran community members in AUD treatment
* Have a primary diagnosis of AUD and are within 30 days of detoxification or last use at time of recruitment

Exclusion Criteria:

* Other medical illnesses that compromise neurocognition
* Active use of prescribed opioids or benzodiazepines that may hinder new learning
* Commitment to complete active phase and attend follow-up
* No pending incarceration or plans to leave the state

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Bell, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Computer Game Play+IDC: Computer arcade games for 13 weeks plus Individual Drug Counseling
  12 computer arcade games for 13 weeks accessed through the same portal as the Cognitive Remediation exercises and formatted similarly.
Period: 13 Week
Arm/Group | CRT+IDC | Computer Game Play+IDC
Started | 29 | 30
Completed | 21 | 16
Not Completed | 8 | 14
Not completed — Lost to Follow-up | 7 | 14
Not completed — Withdrawal by Subject | 1 | 0
Period: 26 Week
Arm/Group | CRT+IDC | Computer Game Play+IDC
Started | 21 | 16
Completed | 16 | 12
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT+IDC | Computer Game Play+IDC | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.79 (9.41) | 54.60 (10.07) | 55.68 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 25 | 29 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 19 | 18 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59
Lifetime Months of Alcohol Use [Mean (Standard Deviation); unit: Months] — Minimum value = 1 month, Maximum value = 1080 months More months of heavy drinking is worse
  Months | 474.07 (190.00) | 436.71 (141.51) | 455.39 (165.76)
Alcohol Use Days in Last 30 Days [Mean (Standard Deviation); unit: Days] — Minimum value is 0 days, Maximum value is 30 days Fewer days is better.
  Days | 5.25 (7.87) | 3.07 (4.93) | 4.14 (6.57)
Alcohol Use Days in Last 90 Days [Mean (Standard Deviation); unit: Days] — Minimum value is 0 days, Maximum value is 90 days Fewer days is better.
  Days | 39.39 (27.13) | 32.24 (23.92) | 35.75 (25.57)
Polysubstance Use Days in the Last 30 Days [Mean (Standard Deviation); unit: Days] — Minimum value is 0 days, Maximum value is 30 days Fewer days is better.
  Days | .73 (2.60) | .42 (1.41) | .57 (2.05)
Polysubstance Use Days in the Last 90 Days [Mean (Standard Deviation); unit: Days] — Minimum value is 0 days, Maximum value is 90 days Fewer days is better.
  Days | 6.22 (16.47) | 6.79 (18.31) | 6.51 (17.39)
Service Connected Disability (Yes) [Count of Participants; unit: Participants] | 7 | 9 | 16
Social Security Disability Income (Yes) [Count of Participants; unit: Participants] | 10 | 6 | 16
Education (years) [Mean (Standard Deviation); unit: years] | 13.31 (1.76) | 13.27 (1.95) | 13.29 (1.84)
Premorbid IQ Estimate (WTAR) [Mean (Standard Deviation); unit: units on a scale] — Minimum score = 60. Maximum = 140 Higher is better
  units on a scale | 100.28 (12.6) | 98.93 (13.3) | 99.61 (12.95)
Overall Neurocognitive Composite Score [Mean (Standard Deviation); unit: T Scores] — 50 indicates the population mean with a standard deviation of 10; Minimum T Score = 30. Maximum = 80; Higher is better
  T Scores | 45.6 (4.8) | 44.3 (6.4) | 44.95 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Days of Heavy Alcohol Use Assessed by Weekly Time Line Follow-back and Breathalyzer
Description: Heavy alcohol use over 90 days as verified by Time Line Follow-back or breathalyzer findings. Minimum = 0. Maximum = 90. Fewer days is better.
Time Frame: 3 months of active treatment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CRT+IDC | Computer Game Play+IDC
Number analyzed (Participants) | 29 | 30
Days | 5.49 (10.85) | 3.0 (5.89)
Statistical Analysis 1: Comparison: CRT+IDC vs Computer Game Play+IDC; Test type: Superiority; p < .05, ANCOVA; covaried for days of heavy drinking over the 30 days prior to randomization; Mean Difference (Final Values) = -2.82, .05% CI 2-sided [-8.23 to 2.588], Standard Error of Mean 2.68

2. Secondary Outcome: Days of Heavy Alcohol Use Assessed by Weekly Time Line Follow-back and Breathalyzer
Description: Days of heavy drinking days over 30 days adjusted for baseline 30 Day heavy drinking days prior to randomization. Minimum = 0. Maximum = 30. Fewer days is better.
Time Frame: 30 days preceding 6 month follow-up, 3 months after active treatment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (Number of Days)
Arm/Group | CRT+IDC | Computer Game Play+IDC
Number analyzed (Participants) | 14 | 11
units on a scale (Number of Days) | 1.67 (1.21) | 1.51 (1.11)
Statistical Analysis 1: Comparison: CRT+IDC vs Computer Game Play+IDC; Test type: Superiority; p < .05, ANCOVA; Days of heavy drinking 30 days prior to randomization; Mean Difference (Final Values) = .16, .05% CI 2-sided [-3.26 to 3.61], Standard Error of Mean 1.66

3. Secondary Outcome: Penn Alcohol Craving Scale
Description: Changes in self-ratings of alcohol craving from baseline to 6 months. Minimum score = 0. Maximum score = 30. Lower is better.
Time Frame: 6 month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CRT+IDC | Computer Game Play+IDC
Number analyzed (Participants) | 29 | 30
score on a scale | 3.94 (1.45) | 4.59 (1.68)
Statistical Analysis 1: Comparison: CRT+IDC vs Computer Game Play+IDC; Test type: Superiority; p = .77, Mixed Models Analysis; Repeated measure with Baseline, 13 weeks and 26 weeks; Mean Difference (Final Values) = 2.94, .05% CI 2-sided [1.45 to 4.43], Standard Error of Mean 1.49

4. Secondary Outcome: Neurocognitive Composite Score (Average of T-scores for Measures of Attention, Processing Speed, Memory, Delayed Recall, Executive Function)
Description: Changes from baseline on Neurocognitive Composite Score Minimum score = 30; Mean = 50 indicates the population mean with a standard deviation of 10; Maximum score = 70. Higher is better.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale (T scores)
Arm/Group | CRT+IDC | Computer Game Play+IDC
Number analyzed (Participants) | 29 | 30
score on a scale (T scores) | 48.15 (1.08) | 46.70 (1.08)
Statistical Analysis 1: Comparison: CRT+IDC vs Computer Game Play+IDC; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-1.61 to 4.50], Standard Error of Mean 1.53

5. Post Hoc Outcome: Clinical Global Index at 6 Months
Description: Clinical Global Index Scale (1 to 7) with 1 being full recovery and total abstinence. Scores 3 and below represent good recovery. Lower scores are better.
Time Frame: 6 months after randomization
Population: Data was extracted from VA medical records and there were many participants who did not have sufficient information in their chart
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CRT+IDC | Computer Game Play+IDC
Number analyzed (Participants) | 10 | 12
units on a scale | 3.00 (1.91) | 3.28 (2.35)
Statistical Analysis 1: Comparison: CRT+IDC vs Computer Game Play+IDC; Test type: Superiority; p = .05, t-test, 2 sided; Mean Difference (Final Values) = 0.46, .05% CI 2-sided [.19 to 1.11], Standard Error of Mean .43

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CRT+IDC | Computer Game Play+IDC
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT+IDC (N=29) | Computer Game Play+IDC (N=30)
Admitted to emergency department for severe alcohol intoxication (Psychiatric disorders) | 0 (0) | 1 (1) — This is a common occurrence in the AUD population and was unrelated to the intervention.

LIMITATIONS AND CAVEATS:
Due to the pandemic, recruitment was below the 90 subjects proposed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT02664038/Prot_SAP_000.pdf